CLINICAL TRIAL: NCT05544435
Title: The Efficacy of Motivational Interviewing on Self-Care Activities in The Management of Type 2 Diabetes Mellitus: The Sample of Turkey
Brief Title: Motivational Interviewing on Self-Care Activities in T2DM: The Sample of Turkey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ETÜ--ULUDAĞ---001
Record Dates: First submitted 2022-09-01; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Motivational İnterviewing; Nursing; Self-caring activities; Turkey
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motivational Interviewing (Experimental): Intervention In addition to the care they always received, MI sessions were conducted by the researcher for the participants in the experimental group. This intervention was conducted as 30-45 minutes of 12 sessions in total for each patient for a period of 3 months by the academic nurse. In these sessions, the agenda was created in accordance with the nature of MI intervention, efforts were made to resolve the ambivalent feelings in the patient, the patient's change phase was determined, the patient's self-confidence for change was determined, it was questioned how much the patient cared for change and the patient was helped in determining the change plan. In addition, during the sessions, the problems patients experienced about self-care activities, the causes of these problems and the barriers in maintaining self-care activities were discussed and efforts were made to create awareness in patients.
  Interventions: Behavioral: Motivational İnterviewing

INTERVENTIONS:
Behavioral: Motivational İnterviewing — Motivational Interviewing (MI), which is one of these methods, is an individual-based counselling approach that can easily be used by nurses who have been trained to help the management of disease in chronic diseases (Berhe et al., 2020; Kızılırmak & Demir, 2018; Maslakpak et al., 2020). The core principles of MI includes expressing empathy by providing acceptance and understanding, realizing inconsistencies, avoiding discussions and supporting self-efficacy (Matinolli et al., 2012). The main purpose of MI is to identify the ambivalent emotions that occur in the patient in health-related activities, to strengthen and encourage insights of patients by supporting healthy lifestyle changes and self-confidence (R.Miller & Rollnick, 2013). Because of its flexibility and ability to be applied in different behavioural aspects, MI can be administered individually and in groups by trained individuals (Maslakpak et al., 2020).

SUMMARY:
Purpose:This study aims to research the effects of motivational interviewing on self-care activities in patients with type 2 diabetes.

Design and Method:This study is a quasi-experimental clinical research with pre-test post-test comparison.12 sessions were held in 3 months in the experimental group with motivational interviewing method.

Findings:After a 3-month follow up, while a significant improvement was observed in post-intervention self-care activities in the experimental group, a significant decrease was observed in all self-care activities except foot care in the control group.

Practice Implications:Motivational interviewing intervention can be used to develop self-care activities in type 2 diabetes patients, especially to guide diabetes nurses.

DETAILED DESCRIPTION:
This study is a quasi-experimental clinical research with pre-test post-test comparison. Population of the study consists of patients who referred to internal medicine outpatient clinic and clinics of a state hospital and who were diagnosed with T2DM between September 2019 and May 2020. The study was initiated with 60 patients who were aged 18 and older, diagnosed with T2DM at least 6 months ago, literate, living in city centre and with a HbA1c value of 6.5% or higher. These patients were described as potential participants by the researchers and experimental (30 patients) and control (30 patients) groups were formed by using simple random numbers table. The participants were explained about the aim of the study and oral and written permissions were taken. During the study period, 6 patients in the experimental group and 3 patients in the control group left the study for various reasons and the study was ended with 51 patients. In data collection, patient information form prepared by the researchers (age, gender, marital status, educational status, disease duration, presence of another chronic disease and smoking status), metabolic variable values (HbA1c and fasting blood sugar) and Summary of diabetes self-care activities scale (SDSCA) developed by Toobert and Glaskow (1994) and revised in 2000 (D.J. Toobert et al., 2000) were used. Summary of diabetes self-care activities scale consists of subscales such as patient diet, exercise, blood sugar test, foot care and smoking. As a result of the calculation of scores, high scores indicate that patients can fulfil self-care behaviors. After the initial data were collected, the patients in the experimental group were given appointments by the researcher for MI intervention. No intervention was performed on the control group participants and they were given appointment for post-test application three months later.

2.1. Intervention In addition to the care they always received, MI sessions were conducted by the researcher for the participants in the experimental group. This intervention was conducted as 30-45 minutes of 12 sessions in total for each patient for a period of 3 months by the academic nurse. In these sessions, the agenda was created in accordance with the nature of MI intervention, efforts were made to resolve the ambivalent feelings in the patient, the patient's change phase was determined, the patient's self-confidence for change was determined, it was questioned how much the patient cared for change and the patient was helped in determining the change plan. In addition, during the sessions, the problems patients experienced about self-care activities, the causes of these problems and the barriers in maintaining self-care activities were discussed and efforts were made to create awareness in patients.

In each MI session;

* Opening and structuring; Meeting, information was given about our role and goals in the study, how much time the investigators have, the role of the counselee and about there will be detailed questions during the study and the session was opened with the question What is on your mind?'
* Creating agenda: What are the investigators going to talk about today? (What would participants like to talk about today, having your blood sugar measured, eating healthily, getting your medication or exercising/Maybe there is something else?)
* Decision balance: Conflict was created in individuals by asking them to compare their existing healthcare behaviors and ideal/desired healthcare behaviors.
* Determining significance and confidence: How important is it for participants to fulfil self-care activities? How much confidence do participants have in yourself about this?
* Change plan: After decision balance was established, its suitability for patients was evaluated, at the end of the session, an action (change) plan was created for the desired behavior change and the session was closed by determining the next interview day-hour.

In the last MI session:

* The session was opened by summarizing the previous interview.
* A general discussion was made on change.
* Individuals' self-care activities were evaluated (The Summary of Diabetes Self-Care)
* Appointment was made from the hospital for individuals to have their glycemic values measured and the values were recorded (glycemic laboratory results).
* Closing.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older
* Diagnosed with T2DM at least six months ago
* To be literate
* Living in the city centre
* HbA1c value of 6.5% or higher
* Speak Turkish.

Exclusion Criteria:

* Having any psychiatric disease and mental problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Summary of diabetes self-care activities scale (SDSCA) | 3 months after the start of the study
  Summary of diabetes self-care activities scale consists of patient diet, exercise, blood sugar test, foot care and smoking.

SECONDARY OUTCOMES:
Metabolic variable values | 3 months after the start of the study
  HbA1c and fasting blood sugar

CONTACTS AND LOCATIONS:
Overall Officials: Elanur Uludağ, Dr., Principal Investigator — Erzurum Technical University
Locations (1):
- Erzurum Technical University Faculty, Erzurum, Turkey (Türkiye)